CLINICAL TRIAL: NCT00346424
Title: Phase 3, Multicenter, Multi-National, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Alfimeprase in Subjects With Occluded Central Venous Access Devices
Brief Title: Safety and Efficacy Study of Alfimeprase in Subjects With Occluded Central Catheters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HA006
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Thrombosis; Venous Thrombosis
Keywords: occluded central catheter; central venous access devices dysfunction; withdrawal occlusion; Thrombosis; Venous thrombosis
MeSH Terms: conditions — Thrombosis; Venous Thrombosis | interventions — alfimeprase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alfimeprase

SUMMARY:
The purpose of the study is to compare the safety and effectiveness of alfimeprase to a placebo in restoring function of occluded central catheters.

DETAILED DESCRIPTION:
Primary Outcomes: The ability to withdraw at least 3 ml of blood and infuse more at least 5 mL of sterile saline through the occluded catheter lumen at 15 minutes after receiving initial instillation of study drug.

Secondary Outcomes:

The ability to withdraw at least 3 mL of blood and infuse at least 5 mL of sterile saline through the occluded catheter lumen at 30 minutes following a single instillation of study drug and at 30 minutes following a second instillation of study drug if patency is not restored within 30 minutes of the first instillation.

Safety:

* Adverse events
* Major bleeding events
* Change in laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Unable to withdraw 3 mL of blood from a central venous access device
* Hemodynamically stable
* Available for follow-up assessments

Exclusion Criteria:

* Inability to infuse at least 2 mL of saline through the catheter
* Catheter placed less than 48 hours prior to detection of occlusion
* Catheter used for hemodialysis of pheresis
* Less than 18 years of age
* Evidence of mechanical or nonthrombotic occlusion
* Receipt of any thrombolytic agent within 24 hours of randomization
* In the opinion of the investigator, subject is at "high risk" for bleeding events of embolic complications, or has a condition for which bleeding constitutes a significant hazard
* Increased risk for drug extravasation
* Pregnant, lactating, or actively menstruating women and women of child-bearing potential who are not using adequate contraceptive precautions (e.g. intrauterine device, oral contraceptives, barrier methods, or other contraception deemed adequate by the investigator)
* Known right-to-left cardiac shunt, patent foramen ovale, or atrial/ventricular septal defect
* Participation in any other study of an investigational device, medication, biologic, or other agent within 30 days before enrollment and until the 30-day follow up visit
* Any other subject feature that in the opinion of the investigator should preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Catheter function restoration at fifteen minutes after initial instillation of study drug. | 15 minutes

SECONDARY OUTCOMES:
Catheter function restoration at 30 minutes after initial instillation of study drug. | 30 minutes
Catheter function restoration at 30 minutes after second dose instillation of study drug if patency was not restored after first dose. | additional 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deitcher, M.D., Study Director — ARCA Biopharma, Inc.
Locations (1):
- Corvallis Clinic, Corvallis, Oregon, United States